CLINICAL TRIAL: NCT03070418
Title: Mini Incision Dynamic Hip Screw Technique
Acronym: MIDHST
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Issa, Abdulhamid Sayed, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Abdulhai's Technique
Record Dates: First submitted 2017-02-18; First posted 2017-03-03 (Actual); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Intratrochontric Fracture
Keywords: DHS; DCS; Boyd and Griffin Classification

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Abdulhai (Experimental): One show man technique, it is the same of AO Dynamic Hip Screw (DHS) technique using 4 holes plate or smaller, in this case it is enough to make just a 3 cm skin incision.
  Interventions: Procedure: Mini Incision Dynamic Hip Screw Technique

INTERVENTIONS:
Procedure: Mini Incision Dynamic Hip Screw Technique — This technique is the same of AO Dynamic Hip Screw (DHS) technique using 4 holes plate or smaller, in this case it is enough to make just a 3 cm skin incision over the guide wire that is inserted parallel to the anteversion wire by using the 135° guide fixed on the T-handle; (step 2-2), and continuing AO technique steps, until step 3-4, for the plate assembling we remove the guide wire, and insert the plate sliding it through the skin cut over the femur shaft under the muscles using the plate for dissection the soft tissue above the bone surface non using any tool as periosteal elevator but the plate itself by holding it from its DHS screw canal and in 180 degree rotation position in axial aspect (transvers aspect) using the plate end for soft tissue gentle dissection over the bone, then turning the plate 180 degree over the bone shaft to the right position and sliding the DHS screw plat canal over the DHS screw using the measuring bar. Two skin stitches are enough.

SUMMARY:
Femoral cervical fractures fixation with DHS plate throw 3 cm incision and minimum surgical trauma.

DETAILED DESCRIPTION:
This technique is the same of AO Dynamic Hip Screw (DHS) technique using 4 holes plate or smaller, in this case it is enough to make just a 3 cm skin incision over the guide wire that is inserted parallel to the anteversion wire by using the 135° guide fixed on the T-handle; (step 2-2), and continuing AO technique steps, until step 3-4, for the plate assembling we remove the guide wire, and insert the plate sliding it through the skin cut over the femur shaft under the muscles using the plate for dissection the soft tissue above the bone surface non using any tool as periosteal elevator but the plate itself by holding it from its DHS screw canal and in 180 degree rotation position in axial aspect (transvers aspect) using the plate end for soft tissue gentle dissection over the bone, then turning the plate 180 degree over the bone shaft to the right position and sliding the DHS screw plat canal over the DHS screw using the measuring bar. Two skin stitches are enough.

Technique

Step 1-reduction

In many cases the traction table is used. The reduction is done on this table and before the patient is draped. Important also is to guarantee smooth access of the image intensifier in both planes; AP and lateral.

Step 2-guide wire insertion

1. The anteversion of the femoral neck is determined with a long K-wire inserted with the blunt end first. An alternative is to use a long, non-threaded K-wire.
2. Under X-ray control, the guide wire is inserted parallel to the anteversion wire by using the 135° guide fixed on the T-handle.

Step 3-screw insertion

1. The length of the screw must be measured/determined with the guide wire. Note that the screw must be 10 mm shorter than the length of the guide wire. The surgeon will deduct 10 mm of the measured length to determine the screw length.
2. Set the triple reamer to 10 mm shorter than the measured length. The hole is drilled over the guide wire.
3. Tapping is only required in young patients with dense bone.
4. For the plate assembling we remove the guide wire, and insert the plate sliding it through the skin cut over the femur shaft under the muscles using the plate for dissection the soft tissue above the bone surface non using any tool as periosteal elevator but the plate itself by holding it from its DHS screw canal and in 180 degree rotation position in axial aspect (transvers aspect) using the plate end for soft tissue gentle dissection over the bone, then turning the plate 180 degree over the bone shaft to the right position.

   * The plate is slid over the wrench.
   * The DHS screw is attached to the coupling wrench.
   * The sleeve is assembled over the wrench.

Step 4-plate fixation

Impact the plate in order to have best contact with the femur. The plate is fixed with conventional 4.5 mm screws:

* Drill bit 3.2 mm with sleeve
* Measuring
* Tap (when no self-tapping screws are used)
* Insertion of screw

ELIGIBILITY:
Inclusion Criteria:

* Patients presented with intertrochanteric hip fractures

Exclusion Criteria:

* not operative patients

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-06; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with post surgical trauma | 12 -14 days for soft tissue healing
  mini incision

SECONDARY OUTCOMES:
Proportion of patients with cosmetic scar | Up to 6 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Sayed Issa's Clinic, Aleppo, Syria

IPD SHARING:
Plan to Share IPD: Yes